CLINICAL TRIAL: NCT05997784
Title: Disrupting Noxious Synergies of Indoor Air Pollutants and Their Impact in Childhood Health and Wellbeing, Using Advanced Intelligent Multisensing
Brief Title: Study of Indoor Air Pollutants and Their Impact in Childhood Health and Wellbeing
Acronym: SynAIR-G
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: National and Kapodistrian University of Athens (Other); Tbilisi State Medical University (Other); University of Manchester (Other); University of Oulu (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL23_0206
Record Dates: First submitted 2023-06-23; First posted 2023-08-18 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-07

CONDITIONS: Asthma in Children; Allergy
Keywords: Air pollution; Asthma; Allergy; Epidemiology; Public health; App; Remote sensors
MeSH Terms: conditions — Hypersensitivity; Asthma; Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Performing lung function tests (spirometry and fraction of exhaled nitric oxide (FeNO)) — Performing lung function tests and FeNO following European Respiratory Society (ERS) standardized guidelines, through the MIR portable spirometer and the NIOX Vero®, respectively.
  Spirometry is performed using a portable spirometer. All manoeuvres are performed according to the American Thoracic Society and European Respiratory Society (ATS/ERS) standards.
  FeNO test is a quick and non-invasive test that is easy for children to do. To take the test, the child have to blow into a handheld device (NIOX Vero®). More in detail, children are asked to inhale ambient air through a nitrogen oxide scrubber to total lung capacity, and then exhale for 10 seconds. The test results are available right away.
Other: Filling of standardized questionnaires — (Baseline, Follow-up, Quality of life and Final) allowing to collect data on sociodemographic characteristics, health outcomes, potential risk factors, lifestyle and living environment.
  Health outcomes will consider general health (general status, infections, allergies), respiratory health (asthma symptoms, diagnosis, control, triggers, medications, etc.), perception of health and well-being.
Other: Using an App on a device — Children will have to answer a daily questionnaire on cell phone, tablet, computer...), with the help of parents/caregivers.
  To encourage children to answer the questions, the questionnaires will be incorporated into a game that will also teach them about environmental challenges and pollutants in Europe.
  There will be a general health questionnaire with 3 questions assessed on a Likert scale.
  The application will also include 2 questions on respiratory health, with Yes/No answers. If the answer is Yes to one of the questions, the intensity of symptoms will be assessed on a visual analog scale from 0 to 100 (0 almost no symptoms and 100 the most intense symptoms imaginable).
Other: Urine sample — On a voluntary basis, a urine sample will be collected, as well.
Other: Sensors and devices will be used to assess air pollutants in classrooms during the survey — * Particulate matter (PM) will be assessed with a counter as a well as a remote sensor (Canarin) .
  * Volatile Organic Compound (VOCs) with a passive sampler (Radiello).
  * Virus and bacteria will be collected with a pump.
  The devices will be attached to the classroom wall.
  In addition, dust pollution will be assessed by collecting dust with a vacuum cleaner in order to assess phthalates (Dimethyl phthalate, diethyl phthalates, Di(2-ethylhexyl) phthalate).

SUMMARY:
The number and types of indoor air pollutants in schools is rising, however little is known about the impact of their potentially synergistic interactions, upon schoolchildren health. Among children, highly susceptible individuals to air pollution include allergy and asthma sufferers, and a low socioeconomic background, however no specific guidance is available.

The Syn-Air-G project will develop a comprehensive and responsive multipollutant monitoring system (in accessible and actionable formats) by constructing and deploying novel but validated and improved sensors of chemical and biological (allergens, microbes) pollutants) and advancing environmentally friendly interventions (including air purifiers). Health: A comprehensive multidisciplinary and exposome approach of health effects of multi-pollution in small children.

DETAILED DESCRIPTION:
Exposure to indoor air pollutants is evidently a critical issue for human health. For the paediatric population, good indoor air quality in the school's environment is an important contributor to the overall and respiratory health, attendance, and academic performance , while poor air quality is associated to a high risk for adverse health outcomes, especially in the vulnerable asthmatic population . Viruses, microbes, allergens, and chemical pollutants exhibit a complex interaction with the human immune system, depending upon several factors such as the age, predisposition (e.g., atopy) and identity of the agent . Pollen exposure increases the risk of viral infections, such as those attributed to rhinoviruses (RVs) and SARS-Cov2 , while viruses and allergens have been shown to interact with pollutants such as ozone (O3) and fine particles (PM2.5), increasing their morbidity effects. Viral infections, especially RVs, impair anti-bacterial innate immune responses , thus affecting the overall microbiome homeostasis.

There are suggestions of potential synergies between different environmental factors, including gas and particulate chemical pollutants, allergens, and viral/microbial species, particularly in the sensitive younger ages, however, such synergies have not been addressed in a real-life epidemiological, systematic, longitudinal study.

The list of indoor air pollutants associated with significant burden on health disorders and increasing social and economic costs, is long and expanding, as current knowledge evolves, on this particular subject. The detrimental effects of air pollution on several health aspects have recently been reviewed. Additionally, a joint statement by the American Thoracic Society (ATS) and the European Respiratory Society (ERS) integrated the latest scientific evidence showing that air pollution affects almost all systems of the human body, including the respiratory, cardiovascular, central nervous, and endocrine systems Studies based on google trend models have shown significant impact of pollutants on respiratory symptoms, especially during increased pollen season in sensitized individuals . Children, one of the most susceptible subgroups in the population, spend a large proportion of their time indoors such as in the school environments, thus, raising the interest in characterizing the health relevant air pollutants in this microenvironment. Studies of air quality composition in classrooms, has shown that several pollutants' levels exceed the recommended air quality standards . The detrimental health effects of exposure to school-derived pollution have been shown for certain pollutants , while a disproportionate effect has been documented in asthmatics, more so in those born prematurely. Schools also act as accumulators of airborne threats, such as viruses or allergens, which are of particular importance to a large but quite vulnerable proportion of the paediatric population: those will allergies and asthma . Allergens are well known elicitors of respiratory symptoms in sensitized individuals, although the allergen effect is person-specific and non-linear , while associations between aeroallergen exposure in schools and increased asthma morbidity has been documented . Although there is evidence suggesting potential synergies between several different factors, health effects of pollutants are more frequently assessed individually, while results on studies assessing multiple pollutants provide divergent results . The cumulative and/or synergistic exposure between chemical and biological (allergens, microbes) pollutants and how these may affect respiratory symptoms, immune, and mental health and DNA damage is barely known. Moreover, school-based environmental interventions on health outcomes studies, are small and not adequately powered.

The SynAir-Child study, within the context of the EU SynAir-G project, is an epidemiological real-life observational study, aiming to assess if there's a possible association and synergy between indoor air pollutant variability and general, respiratory, immune, and mental health outcomes in school children, based on different socioeconomic backgrounds and on different settings, in different Countries.

Previous studies, such as the European SINPHONIE study, the CAMP study on the association Between Allergen Exposure in Inner-City Schools and Asthma Morbidity Among Students, assessed in real-life settings the composition of school air quality and the impact of certain environmental elements on different health outcomes. Although the indication and aim of the studies is similar, the design of the SynAir-Child study provides a unique setting to prospectively assess the synergistic effects of pollutants at school and outdoor on several health aspects in a large and diverse cohort. In addition, outcomes that constitute an adverse health effect of air pollution on humans' health, as stated in the joint ERS/ATS policy statement, will be evaluated and included in the study. Most importantly, the continuous nature of information provided by sentinel devices set in the schools, will provide an individualized baseline of specific indicators that will be monitored during the follow-up period, to identify personalized health alterations, instead of comparing to generalized standards. It is estimated that the use of a personalized physiological profile can more accurately detect subtle changes in an individual's health markers, leading to a greater likelihood of early detection, in relation to the cumulative environmental exposures. Health outcome data, including respiratory health, immune fitness and both mental and non-mental perspectives will contribute to pollution sensing in an iterative way.

ELIGIBILITY:
Inclusion Criteria:

* Child attending CM1 level at the beginning of the school year
* Child in a classroom selected for the project
* Child and caregiver(s) willing to follow the study procedures.

Exclusion Criteria:

Child or child's parents/guardian's who:

* Refuse to participate to the project / to give informed consent
* Do not want to use the application to fill the questionnaire and follow the protocol procedures.
* Do not read or/and write in French
* Plan a long stay outside the region that does not allow them to follow the visit plan

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: A maximum of 500 schoolchildren at CM1 level (French education system), equally distributed between males and females, will derive from a maximum of eight primary schools and 2-3 classes of CM1 in each school, when available. Therefore, two-three classrooms per schools, in no more than 8 schools, each year, over 2 consecutive school years will be monitored, and children will be followed-up during 10 months.
  The selection of schools will be based on socioeconomic and air pollution criteria (differences between different regions of the participating centres) and whenever possible on annual reports on air quality (if available) from the respectively Directorate of Climate Change and Atmospheric Quality of the Ministry of Environment.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Indoor classroom air concentrations of Pollutants and dust | For 10 Months
  Classrooms concentrations (mean with standard deviation SD) of Viruses, Microbe, Allergens, Chemical Air Pollutants (particulate mater PM , NO2, VOCs, phthalates) (ppm part per million) in air and dust.
Prevalence for respiratory disease | For 10 Months
  Health outcomes measures by the prevalence (%) for allergic and respiratory health reported physician-based diagnosis of asthma and/or allergies.
  Questionnaires about respiratory health disease based on validated International Study of Asthma and Allergies in Childhood (ISAAC) and PreDicta respiratory
  * Asthma Control Test (ACT) composed of 7 items with a Score 20 to 25 means a well-controlled asthma, Score 15 - 19: partially controlled asthma and a Score < 15 means an uncontrolled asthma
  * Asthma control questionnaire (ACQ) composed of 7 items and Scores range between 0 (totally controlled asthma) and 6 (severely uncontrolled).)
  * Visual Analogic Scale (VAS) Questionnaire on the App (a score of 0 no symptoms and 100 the most respiratory symptoms)
Association between asthma and indoor air contaminants | For 10 Months
  Significant association of indoor air quality contaminants and their interactions with health outcomes in schoolchildren: odds-ratio and 95% confidence interval between active asthma and indoor air total Volatile Organic Compound (VOCs) and dust phthalates.

SECONDARY OUTCOMES:
prevalence of children presenting airways obstruction | Between baseline and 10 Months
  In children, the severity of airway obstruction can be graded according to Forced expiratory volume in one second (FEV1) measured by spirometry, percentage predicted measured by spirometry: FEV1 <100% to 80% indicates mild obstruction in children; FEV1 <80% to 50% indicates moderate obstruction; FEV1 <50% to 30% indicates severe airway obstruction; and FEV1 <30% indicates very severe obstruction.
Prevalence of children with an abnormal FeNO | Between baseline and 10 Months
  Percentages of children with an abnormal FeNO. In clinical practice, a normal FeNO test in children is any number less than 20 parts per billion (ppb) in patients without lung inflammation.
  The FeNO will be measured with a handheld device (NIOX Vero®).
Quality of life and wellbeing | At 10 months
  General health outcomes will be measured with the use of a subset of questions from the Child Health Questionnaire (CHD) with 13 items, height (centimeter) and weight (kilogram) Quality of life will be measured with the validated Pediatric Quality of Life (PedsQL) questionnaire composed of 23 items and score on a reverse scale of 100 points. ("Never") = 100 = better quality of life, ("Almost Never") = 75("Sometimes") = 50("Often") = 25 ("Almost Always") = 0 = worst quality of life.
diagnosis of any disease and respiratory diseases | At 10 months
  General health confirmed by questionnaire and physicians based diagnosis VAS Questionnaire on the app Through Quality of life and wellbeing questionnaires based on validated International Study of Asthma and Allergies in Childhood (ISAAC), PreDicta respiratory, ACT, ACQ
Environmental source of pollutants | Baseline
  Children and their caregivers will answer standardized questionnaires on sources and exposures of pollutant. (qualitative questionnaire, no scoring)

CONTACTS AND LOCATIONS:
Overall Officials: Davide CAIMMI, CAIMMI, Study Director — CHU de Montpellier
Locations (1):
- University Hospital of Montpellier, Montpellier, Occitanie, France

IPD SHARING:
Plan to Share IPD: Undecided